CLINICAL TRIAL: NCT00483912
Title: Molecular Adsorbent Recirculating System (MARS) in Severe Acute Pancreatitis
Brief Title: Albumindialysis in Acute Pancreatitis
Acronym: pancreatitis
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: R04005
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2007-06-08 (Estimated); Status verified 2007-06

CONDITIONS: Pancreatitis; Multiple Organ Failure
Keywords: pancreatitis, MARS; severe acute pancreatitis with early multiple organ failure
MeSH Terms: conditions — Pancreatitis; Multiple Organ Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Molecular adsorbent recirculating system

SUMMARY:
The incidence of acute pancreatitis has been doubled during last three decades in Finland. Alcohol is the main cause of acute pancreatitis in Finland accounting for 70 % of cases. Although the mortality of acute pancreatitis has been decreased it still appears and especially early multiple organ failure is the main cause of all deaths. Multiple organ failure in the early course of the disease is thought to be caused by the release of cytokines. Molecular adsorbent recirculating system (MARS) has shown to decrease mortality in acute alcohol hepatitis and paracetamol intoxication. Also it has been shown to improve kidney function due to hypoperfusion and tubulus necrosis and overrule decrease mortality in patients with multiple organ failure due to different reasons. A part of patients with acute alcoholic pancreatitis may have so-called fat liver already on admission. It has been shown that the highest mortality is especially associated those with early liver and kidney failure. MARS treatment has never earlier been used in the patients with acute alcoholic pancreatitis and early organ failure. In this study we randomize patients with acute alcoholic pancreatitis and early multiple organ failure (Sofa score>2) to two groups: 1) Standard pancreatitis treatment in intensive care unit and 2) Standard pancreatitis treatment in intensive care unit with 5 MARS sessions.

ELIGIBILITY:
Inclusion Criteria:

* Severe acute alcoholic pancreatitis with early multiple organ failure (Sofa score >2)

Exclusion Criteria:

* If patient or his/her family member refuses, pregnancy.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Sari Räty, Study Chair — Dept. of Gastroenterology and Alimentary Tract Surgery
Locations (1):
- Tampere University Hospital, Tampere, Finland